CLINICAL TRIAL: NCT01631149
Title: Effect of Deep BLock on Intraoperative Surgical Conditions, Perioperative Hemodynamic Status and Respiratory Parameters Following Reversal With Sugammadex in Patients Undergoing Laparoscopic Renal and Prostate Surgery.
Brief Title: Effect of Deep BLock on Intraoperative Surgical Conditions
Acronym: BLISS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Albert Dahan, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: bliss s
Record Dates: First submitted 2012-06-19; First posted 2012-06-28 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Hypertrophy; Renal Disease
Keywords: urology; muscle relaxation; laparoscopy; anesthesia; rocuronium
MeSH Terms: conditions — Prostatic Hyperplasia; Kidney Diseases | interventions — Rocuronium; Atracurium; Mivacurium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep surgical block (Experimental): Continuous rocuronium infusion will be used to induce a deep surgical block with post tetanic twitch count of max 2. Rocuronium loading dose = 1.0 mg/kg, followed by 0.6-1.0 mg/kg per hour.
  Interventions: Drug: Surgical block (rocuronium; atracurium/mivacurium)
- Moderate/normal surgical block (Active Comparator): A normal block will be induced by an atracurium bolus dose followed by a mivacurium infusion to induce a train of four count of 1-2.
  Interventions: Drug: Surgical block (rocuronium; atracurium/mivacurium)

INTERVENTIONS:
Drug: Surgical block (rocuronium; atracurium/mivacurium) — The surgical block will be varied by either induction of a deep block (via rocuronium infusion) or a moderate/normal block (using atracurium/mivacurium infusion)
  Other Names: deep muscle blockade
  Arms: Deep surgical block
Drug: Surgical block (rocuronium; atracurium/mivacurium) — A surgical block will be induced by infusion of either rocuronium (deep block) or atracurium/mivacurium (normal/moderate block)
  Other Names: moderate muscle blockade
  Arms: Moderate/normal surgical block

SUMMARY:
Rationale: A deep neuromuscular block is often associated with improved surgical conditions especially in laparoscopic surgery. However, a deep block comes at the expense of a variety of items that may conflict with the use of a deep surgical muscle blockade including a long recovery phase, the need for muscle reversal, postoperative ventilation, impaired postoperative breathing. With the introduction of Sugammadex there is now the possibility to reverse an even deep surgical block. This may overcome most if not all of the issues mentioned.

Objective: To assess whether a deep neuromuscular block provides better surgical conditions than a moderately deep block as derived from a surgical rating score.

Study design: Single center, double-blind randomized controlled trial. Study population: 24 ASA I-III patients scheduled for laparoscopic renal (n=12, GROUP 1) or prostatic surgery (n=12, GROUP 2).

Intervention: In both GROUP 1 and GROUP 2, 6 six patients will receive neuromuscular blockade according to current practice (atracurium (bolus) plus mivacurium (cont. infusion)) aimed at a moderately deep neuromuscular block (1-2 twitches in the Train of Four (TOF) monitor). The other six will receive a bolus plus continuous infusion with rocuronium aimed at a deep neuromuscular block (1-2 twitches post tetanic count (PTC)). All surgical procedures will be performed by one surgeon.

Main study parameters/endpoints: To study the surgical conditions in patients undergoing laparoscopic renal or prostate surgery during deep versus less deep neuromuscular block as assessed by the surgical rating score.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Compared to current practice there will be no additional risk.

DETAILED DESCRIPTION:
Surgical conditions in laparoscopic surgery are largely determined by the degree of neuromuscular relaxation during surgery. Especially in procedures which are confined to a narrow working field such as renal and prostatic laparoscopic surgery, deep neuromuscular relaxation may be beneficial. Until recently however, deep neuromuscular block (1-2 twitches post tetanic count) came at the expense of a variety of items that conflicted with its use. Occurrence of postoperative residual neuromuscular blockade after deep neuromuscular block was a common adverse event. Residual neuromuscular block is a risk factor for developing airway obstruction and pulmonary complications such pneumonia and atelectasis. The use of acetylcholinesterase inhibitors, like neostigmine, as a traditional neuromuscular blocking reversal agent, have a slow onset of action. Side effects due to muscarine receptor stimulation are bradycardia, hypersalivation, nausea and vomiting. Coadministration of a muscarine agonist like atropine is often necessary to address the heart rate-related side effects of neostigmine. Atropine, however, in itself may induce other side effects.

Rapid, safe and complete reversal of neuromuscular blockade was not possible until the discovery of Sugammadex. Sugammadex is a modified y-cyclodextrin. It was developed to selectively bind free plasma rocuronium, a non-depolarizing steroidal neuromuscular blocking agent. By binding free rocuronium, less rocuronium becomes available at the neuromuscular junction to bind to the muscarine receptor. Non-depolarizing neuromuscular blocking agents (NMBA's) block the muscarine receptor at the neuromuscular junction, making them unavailable to acetylcholine based signal transmission. Sugammadex has proven to rapidly and safely reverse rocuronium and vecuronium. Even high dose rocuronium (1.2 mg/kg and continuous rocuronium infusion used to achieve deep neuromuscular blockade can safely be reversed by Sugammadex.

Theoretically, the availability of Sugammadex makes it possible to use deep neuromuscular block (DNB) during surgery to improve surgical conditions without the occurrence of the above-mentioned adverse events. The use of DNB to improve surgical conditions, however, has not yet been evaluated. The investigators therefore aim to investigate the use of rocuronium induced-DNB in renal and prostatic laparoscopic surgery. Current anesthesiologic practice during these procedures in the LUMC consists of an intravenous (propofol) or volatile (sevoflurane) anesthetic combined with mivacurium and atracurium to achieve a moderately deep neuromuscular block (0-2 twitches TOF). Reversal of NMB is by the neostigmine atropine combination. In the current study the investigators will assess the effect of a DNB (1-2 twitches post tetanic count) using a continuous rocuronium infusion on surgical conditions. After surgery Sugammadex 4 mg/kg will be used to safely and rapidly reverse the neuromuscular blockade within 5-min.

The main end-point of the study is the effect of the deep block on the surgical conditions. The investigators will study these conditions using two methods. (1) Assessment of the surgical condition by the operating surgeon (all surgeries will be performed by one surgeon), using a 5-point rating surgical rating scale from 1 (= extremely poor surgical condition) to 5 = optimal surgical condition. (2) Video images, used by the surgeon to perform the surgery, will be rated by a team of surgical and non-surgical experts. Apart from the additional scoring data, this approach allows for the validation of the surgical rating scale.

Minor end-points of the study are (1) measurement of hemodynamics during surgery using a non-invasive cardiac output and blood pressure device. Assuming that intra-abdominal pressure will affect the venous return and hence cardiac output during surgery, a deep neuromuscular block might affect the hemodynamic parameters positively; (2) measurement of respiration, pain, and alertness in the recovery room to assess whether reversal with Sugammadex influences these parameters positively compared to neostigmine/atropine reversal.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with renal or prostatic disease who are will undergo an elective laparoscopic renal surgical procedure or laparoscopic prostatectomy;
* ASA class I-III
* > 18 years of age;
* Ability to give oral and written informed consent

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing neuromuscular function;
* Allergies to muscle relaxants, anesthetics or narcotics;
* A (family) history of malignant hyperthermia;
* Patients who have a contraindication for neostigmine administration;
* Women who are or may be pregnant or are currently breast feeding;
* Renal insufficiency, as defined by serum creatinine x 2 of normal, or urine output < 0.5 ml/kg/h for at least 6 h. When available, other indices will be taken into account as well such as glomerular filtration rate < 60 ml/h and proteinuria (a ratio of 30 mg albumin to 1 g of creatinine).
* Previous retroperitoneal surgery at the site of the current surgery.
* Body mass index > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD {hD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boon M, Martini CH, Aarts LP, Bevers RF, Dahan A. Effect of variations in depth of neuromuscular blockade on rating of surgical conditions by surgeon and anesthesiologist in patients undergoing laparoscopic renal or prostatic surgery (BLISS trial): study protocol for a randomized controlled trial. Trials. 2013 Mar 1;14:63. doi: 10.1186/1745-6215-14-63. PMID 23452344
- See also: Website of the hospital in which the study will be performed — http://www.lumc.nl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 patients were recruited. In 4 one or more exclusion criteria were met, the others were randomized; 2 patients withdrew consent; two others replaced them.
Pre-assignment Details: No significant events occurred that delayed or interfered with the enrollment
Period: Overall Study
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 60 (12) | 60 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Netherlands | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Surgical Rating Scale
Description: During the procedure, the surgical condition will be scored by the surgeon using a 5-point surgical rating scale. In order to reduce variability in the surgical rating all surgeries will be performed by one single surgeon. The rating scale will be a 5-point ordinal scale ranging from 1 = poor condition to 5 = optimal surgical conditions. The surgeon will score the condition at 15 minute intervals. In case of a sudden change in surgical conditions additional scores will be added to the case record form. If conditions are poor (score 1 or 2), muscle relaxation will be increased, a score of 1 will be used.
  In each subject the scores over time were averaged and a comparison between treatments was performed using a t-test
Time Frame: Measurements will be made during the stay in the operating room for an average period of 3 hours
Population: Each participant that was dosed was analyzed
Measure: Mean (Standard Deviation); unit: units on a scale (1-5)
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block
Number analyzed (Participants) | 12 | 12
units on a scale (1-5) | 4 (0.4) | 4.7 (0.4)
Statistical Analysis 1: Comparison: Moderate/Normal Surgical Block vs Deep Surgical Block; The individual scores obtained during surgery were averaged. The average values were compared using a t-test between treatments; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.7, Standard Deviation 0.4

2. Secondary Outcome: Breathing
Description: In the recovery room the respiratory rate will be measured continuously using the Respir8 respiratory rate monitor. The data will be recorded on the CRF at 15 min intervals.
  Breathing rate units are "number of breaths" as measured in 1 min.
  Comparison by t-test: NS between treatments
Time Frame: Measurements will be made during the stay in the recovery room for an average period of 3 hours
Population: In each subject the scores over time were averaged and a comparison between treatments was performed using a t-test
Measure: Mean (Standard Deviation); unit: breaths per min
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block
Number analyzed (Participants) | 12 | 12
breaths per min | 14.5 (2.2) | 14.5 (2.2)

3. Secondary Outcome: Post-operative Pain
Description: Using a 10 cm visual analogue score pain relief score will be measured. 0 = no pain 10 = most severe pain
  No statistical analysis was performed!
Time Frame: measurements are made in the recovery room following surgery for an average prior of 1 hour
Population: The pain data were averaged over time and compared by t-test between groups
Measure: Mean (Standard Deviation); unit: units on a scale (0-10 cm)
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block
Number analyzed (Participants) | 12 | 12
units on a scale (0-10 cm) | 2.6 (1.6) | 2.1 (2.2)

4. Secondary Outcome: Postoperative Sedation Score
Description: Using a 5-point sedation scale, sedation levels will be obtained throughout the postoperative period.
  0 = wide awake 5= severely sedated, The sedation data were averaged over time.
Time Frame: Measurements will be made during the stay in the operating room for an average period of 3 hours
Measure: Mean (Standard Error); unit: units on a scale (0-5)
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block
Number analyzed (Participants) | 12 | 12
units on a scale (0-5) | 2.0 (0.6) | 1.3 (1.0)

5. Secondary Outcome: Nausea and Vomiting
Description: Using a yes - no questionnaire, the patients will be asked whether they are nauseated or not or whether they vomited. In fact yes indicates the nr of participants.
  No statistical analysis was performed.
Time Frame: Measurements will be made during the stay in the operating room for an average period of 3 hours
Measure: Number; unit: participants
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 4-5 hours
Arm/Group | Moderate/Normal Surgical Block | Deep Surgical Block
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No